CLINICAL TRIAL: NCT02771444
Title: Low Dose Tomosynthesis Compared to Traditional Tomosynthesis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Decision by sponsor, development stopped.
Sponsor: Philips Digital Mammography Sweden AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DOC-EMOA-A7UDZ2
Record Dates: First submitted 2016-05-10; First posted 2016-05-13 (Estimated); Last update posted 2018-03-26 (Actual); Status verified 2018-01

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Masking Description: This is an imaging study. All participants will be imaged using two modalities. All participant data will be deidentified.
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tomo Assessment (Experimental): Subjects will have a 4-view tomosynthesis examination with the study device.
  Interventions: Device: Tomo Assessment

INTERVENTIONS:
Device: Tomo Assessment — A four-view tomosynthesis examination
  Other Names: MicroDose Tomosynthesis

SUMMARY:
This study aims to evaluate image quality of a low-dose tomosynthesis system versus a comparator. Subjects will undergo a four-view tomosynthesis examination with the comparator and with the study device, and images will be assessed by several radiologists by comparing details in the images from the two systems.

DETAILED DESCRIPTION:
Tomosynthesis is a relatively new technology to acquire mammographic images where images are acquired over several projection angles, giving 3d information that can help radiologists assess images.

The aim of the study is to see whether a new low-dose tomosynthesis system has comparable image quality at a lower x-ray radiation dose to a comparator.

ELIGIBILITY:
Inclusion Criteria:

* Woman over 40 years of age
* Has a tomosynthesis examination with comparator
* Has a mammographic finding

Exclusion Criteria:

* Pregnant, breastfeeding or believes she may be pregnant
* Unable or unwilling to give informed consent

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2018-03-22 (Actual); Study Completion 2018-03-22 (Actual)

PRIMARY OUTCOMES:
X-ray dose | 4 months
  X-ray dose will be measured per projection.

SECONDARY OUTCOMES:
Lesion conspicuity comparison of images from study device vs comparator | 4 months
  Lesion conspicuity will be assessed by image readers (radiologists) comparing the conspicuity of the same lesion imaged with the study device to the comparator

CONTACTS AND LOCATIONS:
Overall Officials: Pietro Panizza, M.D, Principal Investigator — Ospedale San Raffaele
Locations (1):
- Ospedale San Rafaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Venturini E, Losio C, Rodighiero M, Ferrarese G, Del Vecchio A, Loria A, Rehn JR, Panizza P. Low dose photon-counting digital breast tomosynthesis: comparison with a commercially available tomosynthesis unit in the detection and characterization of breast carcinomas. Radiol Med. 2025 Oct 4. doi: 10.1007/s11547-025-02115-7. Online ahead of print. PMID 41045355